CLINICAL TRIAL: NCT05203601
Title: A Phase Ⅰa Clinical Study Exploring Safety, Tolerability, Pharmacokinetics, Immunogenicity and Preliminary Efficacy of SIBP-03 When Treating the Patients With Advanced Malignant Solid Tumors.
Brief Title: A Phase Ⅰa Clinical Study Exploring Efficacy of SIBP-03 When Treating the Patients With Advanced Malignant Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SIBP-03-01
Record Dates: First submitted 2022-01-06; First posted 2022-01-24 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Tumor
Keywords: Monoclonal antibody; HER3; safety; efficacy; pharmacokinetics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a dose escalation and extension study which designed as an open and multi-dose escalation study with single and multiple dosing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIBP-03(Recombinant anti-HER3 humanized monoclonal antibody injection) (Experimental): Stage 1: dose escalation stage Injection, first dose 2mg/kg, then 5mg/kg until the dose are no longer met the requirements of continuing the trial or up to 40 mg/kg.
  Stage 2: joint extension stage:
  ① Group of advanced head and neck squamous cell carcinoma ：SIBP-03 & Cetuximab 5mg/kg dose level: Sibp-03, 5 mg/kg, Q3W Cetuximab, 400 mg/m2 (week 1), 250 mg/m2 (weekly follow-up), QW 10mg/kg dose level: Sibp-03, 10 mg/kg, q3W Cetuximab, 400 mg/m2 (week 1), 250 mg/m2 (weekly follow-up), QW
  ② Group of breast cancer：SIBP-03 & Trastuzumab & Docetaxel 5mg/kg dose level: Sibp-03, 5 mg/kg, Q3W Trastuzumab, first dose 8 mg/kg, maintenance dose 6 mg/kg, q3w+ Docetaxel 75mg/m2 q3w.
  10mg/kg dose level: Sibp-03, 10 mg/kg, q3W Trastuzumab, first dose 8 mg/kg, maintenance dose 6 mg/kg, q3w+ Docetaxel 75mg/m2 q3w.
  Interventions: Biological: SIBP-03

INTERVENTIONS:
Biological: SIBP-03 — Stage 1:
  Six dose groups of 2, 5, 10, 15, 20 and 40 mg/kg were planned. Dose increments began at 2 mg/kg using accelerated titration. In the first dose group, after the first patient was injected with Sibp-03, if the subject developed toxicity grade ≥2（CTCAE v5.0 standard）within 21 days of initial administration，then the subject increased to 3 and the study design method in this dose level convert to "3+3". If the subject didn't develop toxicity grade ≥2, then the study of the second and next dose group can be carried out using "3+3" incremental design.
  Stage 2:
  Cohort 1 included patients with advanced head and neck squamous cell carcinoma and cohort 2 included patients with breast cancer. According to the results of dose escalation stage and similar drug trials, 5mg/kg and 10mg/kg dose levels were selected to enter this phase. Each cohort will be extended to include 6-8 subjects to receive this product in combination with the standard treatment study.

SUMMARY:
The main purpose of

• To evaluate the safety, tolerability and pharmacokinetic characteristics of SIBP-03（Recombinant anti-HER3 humanized monoclonal antibody injection）.

A secondary purpose

* Assess the immunogenicity of SIBP-03. Exploratory purpose
* Explore potential biomarkers;
* Preliminary evaluation of the antitumor efficacy of SIBP-03.

DETAILED DESCRIPTION:
To evaluate the safety, tolerability, pharmacokinetics, immunogenicity and preliminary efficacy of recombinant anti-HER3 humanized monoclonal antibody injection when treating the patients with advanced malignant solid tumors. This study is an open, multi-dose escalation and extension study of single and multiple dosing. This study was divided into two phases: the first phase was dose escalation phase, the second phase was joint expansion phase, in which the dose escalation phase was a single-center study, and the joint expansion phase was a multi-center study. Stage 1, dose escalation stage: Six dose groups of 2, 5, 10, 15, 20 and 40 mg/kg were planned, then exploring the most appropriate dose. The second stage, combined use extension stage: According to the preliminary data of drug safety, tolerance, pharmacokinetics and efficacy obtained in the dose escalation stage, combined with the clinical study results of similar drugs, 5mg/kg and 10mg/kg dose levels were selected to enter the combined extension stage and used in patients with advanced head and neck squamous cell carcinoma or with breast cancer.

ELIGIBILITY:
The inclusion criteria:

* Male and female aged between 18 and 75 years old.
* The enrolled subjects shall conform to the following criteria (Dose Escalation phase): Histologically or cytologically confirmed locally advanced or metastatic solid tumours resistant or refractory to conventional treatment, for which no conventional therapy exists or is not considered appropriate by the Investigator. (Priority for inclusion but not limited to head and neck squamous cell carcinoma, esophageal squamous cell carcinoma and breast cancer with high HER2 expression).
* The enrolled subjects shall conform to the following criteria (Joint extension phase): Cohort 1: Patients in recurrent/metastatic advanced head and neck squamous cell carcinoma (HNSCC) who is histologically or cytologically confirmed. The patient is also unsuitable for radical surgical resection, failed from standard treatment, or previously treated by PD-1 mAb therapy (unless patient is not suitable for PD-1 therapy). Cohort 2: Patients in advanced breast cancer (BC) with her2-overexpression who is histopathologically or cytologically confirmed, previously untreated with anti-HER2-targeted therapy such as trastuzumab or eligible for re-use though once been treated with trastuzumab.
* At least one targeted lesion that is measurable (according to RECIST V1.1 criteria, CT or MRI) and that lesion has not received radiation therapy.
* ECOG fitness score is between 0 and 1.
* Life expectancy of at least 3 mouths.
* Adequate organ function（No blood transfusion, granulocyte colony-stimulating factor (G-CSF injection, or other medical support within 14 days prior to the use of the investigational drug)
* The blood pregnancy test for women of reproductive age was negative during the screening period, and subjects of reproductive age (including male subjects) have no pregnancy plan and shall voluntarily use effective contraception during the trial and 6 months after the last dose.
* Voluntarily participate in this study and provide written informed consent.

The exclusion criteria:

* Subjects with the following tumors: Malignancy other than the tumor treated in this study during the past 5 years (except for thyroid cancer, cured basal cell carcinoma of the skin, and carcinoma in situ of the cervix). Untreated central nervous system (CNS) primary tumors or metastases. Meningeal metastatic carcinoma. Patients with BMS who had previously received systemic and radical BMS treatment (radiotherapy or surgery), and who had been stable without any clinical symptoms for at least 4 weeks with systemic hormone therapy been stopped for more than 2 weeks.
* Subjects who have any of the following treatment history or surgical history, or who plan to receive any of the following antitumor treatments during the trial period： Patients who received proprietary Chinese medicines whose specifications explicitly included antitumor effects within 2 weeks prior to the first dose. Patients undergoing maintenance therapy within 6 months after surgery. Patients who have not recovered to normal or ≤level 1 toxicity from previous treatment (except for hair loss). Patients who received major surgery, radiation, biotherapy, or chemotherapy within 4 weeks prior to initial dose, or who were systematically treated by other investigational agents with unhealed surgical wounds, ulcers or fractures. Patients scheduled to receive any other antitumor therapy during the trial period should be excluded (except for testosterone reduction therapy in prostate cancer patients). Patients received immunosuppressants or any systemic corticosteroids within 1 week prior to the first dose. Patients previously treated with anti-HER3 drug.
* The subject's past medical history or laboratory examination shows any of the following abnormalities: Abnormal coagulation function with bleeding tendency or receiving thrombolytic or anticoagulant therapy or with blood loss/donation of more than 200 mL within 2 months prior to drug administration. A history of immunodeficiency, including positive HIV, or other acquired or congenital immunodeficiency disease, or a history of organ transplantation. A past history of neurological or psychiatric disorders, including epilepsy or dementia.
* Patients with positive TP test during screening period; with active HBV、HCV infection; except for stable hepatitis B infection by drug therapy (DNA titer not higher than 500 IU/mL or copy number <1000 copies/mL) and cured hepatitis C infection(negative HCV RNA test).
* Ascites, pleural effusion and pericardial effusion with clinical symptoms during the screening period, or patients requiring drainage or previously drained within 4 weeks prior to initial dose.
* Concommitted with a serious, progressive, or uncontrolled illness, assessed by the investigator to increase the risk of study participation during the screening period, including but not limited to: Cerebrovascular accident or transient ischemic attack (within 6 months prior to screening). Heart disease judged by the investigator to be unsuitable for the study, abnormal cardiac function or renal function with severity≥grade II.
* Concomitant diseases (e.g. severe hypertension, diabetes, thyroid disease, active infection, etc.) that seriously endanger patients' safety or affect patients' ability to complete the study, according to the investigator's judgment.
* Have a history of severe allergy, or allergic to protein products, CHO cell products, other recombinant human or humanized antibodies or components of the investigational drug.
* Female who is pregnant or lactating.
* Patients deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
AE(Adverse Events) | 28 days after the last dose
  That is adverse events, any adverse events that occurred to the subject during the study period.
SAE(Serious Adverse Events) | 28 days after the last dose
  That is serious adverse events, any serious adverse events that occurred to the subject during the study period.
AUC(Area Under The Plasma Concentration Versus Time Curve) | 28 days after the last dose
  It shows the degree to which a drug is absorbed and used in the body.
Cmax(Peak Plasma Concentration) | 28 days after the last dose
  It shows the highest plasma concentration of a drug that can be achieved after administration
Tmax(Peak Time) | 28 days after the last dose
  That is peak time of drug action, it shows the time required to reach the maximum concentration on the subject plasma concentration curve after administration.
T ½（Terminal elimination half-life） | 28 days after the last dose
  It reflects how quickly the drug is eliminated from the body.
CL（Clearance Rate） | 28 days after the last dose
  Apparent volume of drug distribution removed from the body per unit time.
Pulse rate | 28 days after the last dose
  Pulse rate of the subject.
Respiratory rate | 28 days after the last dose
  Respiratory rate of the subject.
Body temperature | 28 days after the last dose
  Body temperature of the subject.
Blood pressure | 28 days after the last dose
  Blood pressure of the subject.

SECONDARY OUTCOMES:
ADA(Anti-drug Antibody) | The 1 day the test results reported after the last dose
  The incidence of anti-drug antibody.
NAb(Neutralizing Antibody) | The 1 day the test results reported after the last dose
  The incidence of neutralizing antibody.

OTHER OUTCOMES:
ORR(Objective Response Rate) | The 1 day the test results reported after the last dose
  The proportion of subjects whose tumor volume shrinks to a predetermined value and maintains the minimum time limit, and is the sum of complete and partial responses.
DCR(Disease control rate) | The 1 day the test results reported after the last dose
  In clinical trials, the percentage of subjects with advanced or metastatic cancer who responded fully to cancer treatment, partially responded, and had stable disease .
PFS(Progression-free survival) | The 1 day the test results reported after the last dose
  The time between the onset of randomization and the onset (of any aspect) of tumor progression or death (from any cause).
HER3 in the blood | The 1 day the test results reported after the last dose
  A protein in the blood.
NRG1 in the blood | The 1 day the test results reported after the last dose
  A protein in the blood.
Her2 | The 1 day the test results reported after the last dose
  A protein in pathological tissues.
Her3 in pathological tissues | The 1 day the test results reported after the last dose
  A protein in pathological tissues.
NRG1 in pathological tissues | The 1 day the test results reported after the last dose
  A protein in pathological tissues.
EGFR(protein) | The 1 day the test results reported after the last dose
  A protein in pathological tissues.
FAT1 | The 1 day the test results reported after the last dose
  A gene in pathological tissues.
Notch1 | The 1 day the test results reported after the last dose
  A gene in pathological tissues.
Notch2 | The 1 day the test results reported after the last dose
  A gene in pathological tissues.
Notc3 | The 1 day the test results reported after the last dose
  A gene in pathological tissues.
Notch4 | The 1 day the test results reported after the last dose
  A gene in pathological tissues.
TP53 | The 1 day the test results reported after the last dose
  A gene in pathological tissues.
PIK3CA | The 1 day the test results reported after the last dose
  A gene in pathological tissues.
EGFR(gene) | The 1 day the test results reported after the last dose
  A gene in pathological tissues.

CONTACTS AND LOCATIONS:
Overall Officials: Co., Ltd Shanghai Institute Of Biological Products, Study Director — Shanghai Institute Of Biological Products; Shanghai Cancer Center Fudan University, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No